CLINICAL TRIAL: NCT05168358
Title: Effect of Overnight Bladder Drainage on Posterior Urethral Valve Sequelae: A Randomized Controlled Trial
Brief Title: Overnight Bladder Drainage and Posterior Urethral Valve Sequelae
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Elkashef, Ahmed Elkashef, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCD-PUV
Record Dates: First submitted 2021-12-12; First posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Posterior Urethral Valve
Keywords: Overnight Catheter Drainage; Posterior Urethral Valve; Randomized Controlled Trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): This arm will include 55 patients, their parents will be taught the timed voiding regimen every 2 hours.
- OCD group (Experimental): This arm will include 55 patients, their parents will be taught the timed voiding regimen every 2 hours, in addition to placing an overnight catheter to drain the urinary bladder during night.
  Interventions: Procedure: Overnight Bladder Drainage

INTERVENTIONS:
Procedure: Overnight Bladder Drainage — Parents or caregivers of the patients will be taught to place an indwelling catheter in the bladder at bedtime for about 8-12 h under a clean technique every night for one year. The catheter will then be allowed to drain freely into a gravity drainage collecting bag or in the diapers. On the next morning, the catheter will be removed and the timed voiding regimen will be resumed.
  Other Names: Overnight Catheter Drainage
  Arms: OCD group

SUMMARY:
We hypothesize that overnight catheter drainage (OCD) of the urinary bladder might improve bladder dynamics and subsequently lead to improvement or resolution of hydronephrosis (HN) and renal function in boys who underwent PUV ablation.

Patients who have persistent HN and bladder dysfunction at least one year after PUV ablation will be randomly allocated into two groups: the first group (control group): 55 patients, their parents will be taught the timed voiding regimen every 2 hours, while the second group (OCD group): 55 patients, their parents will be taught the timed voiding regimen every 2 hours, in addition to placing an overnight catheter to drain the urinary bladder during night.

We will study the effect of OCD of the urinary bladder on the improvement or resolution of HN and urinary bladder function within a year of starting this regimen.

DETAILED DESCRIPTION:
Posterior urethral valve (PUV) is the most common cause of bladder outlet obstruction (BOO) in boys. PUV induces damage to the smooth muscles of the bladder and ureter with subsequent damage to the renal parenchyma. All these sequelae begin antenatally and persist even after successful valve ablation.

The standard management of these sequelae includes timed voiding, double voiding, clean intermittent catheterization (CIC) to facilitate bladder emptying and anticholinergic drugs to improve poor bladder compliance. However, in some polyuric cases even voiding or catheterization as frequently as every 2 hours is not effective to maintain safe bladder volumes especially at night.

Overnight catheter drainage (OCD) of the urinary bladder has been increasingly suggested to be beneficial in protecting the upper tracts of patients with high urine output, defective and poorly compliant bladders, thus resulting in improvement of the renal function, hydronephrosis (HN) and the urodynamic changes as well.

Therefore, we hypothesize that OCD of the urinary bladder might improve bladder dynamics and subsequently lead to improvement or resolution of HN and renal function in boys who underwent PUV ablation.

Patients who have persistent HN and bladder dysfunction at least one year after PUV ablation will be randomly allocated into two groups: the first group (control group): 55 patients, their parents will be taught the timed voiding regimen every 2 hours, while the second group (OCD group): 55 patients, their parents will be taught the timed voiding regimen every 2 hours, in addition to placing an overnight catheter to drain the urinary bladder during night.

We will study the effect of OCD of the urinary bladder on the improvement or resolution of HN and urinary bladder function within a year of starting this regimen by laboratory tests, renal and bladder ultrasonography (US), voiding cystourethrogram (VCUG) and dimercaptosuccinic acid (DMSA) scan. The bladder dynamics will also be examined by urodynamic study (UDS).

ELIGIBILITY:
Inclusion Criteria: Patients who have;

* Persistent hydronephrosis and
* Unfavorable bladder dynamics on urodynamic study performed at least one year after posterior urethral valve ablation will be included in the study. The unfavorable bladder dynamics will be defined as poor compliance or detrusor overactivity.

Exclusion Criteria: Patients who;

* Underwent urinary diversion (e.g. vesicostomy or ureterostomy),
* Have other conditions that could affect lower urinary tract function,
* Have infravesical obstruction or
* Those who will refuse to participate in the study will be excluded.

Ages: 1 Year to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 55 (Estimated)
Dates: Start 2021-12-12 (Actual); Primary Completion 2022-12-12 (Estimated); Study Completion 2023-06-12 (Estimated)

PRIMARY OUTCOMES:
Improvement or Resolution of Hydronephrosis | One Year
  Impact of overnight bladder drainage on improvement or resolution of hydronephrosis assessed by renal and bladder ultrasonography. Improvement of hydronephrosis will be defined as downgrading of hydronephrosis according to Society of Fetal Urology grading system.

SECONDARY OUTCOMES:
Improvement of Bladder and Renal Function and Resolution of Urinary Tract Infection | One Year
  Impact of overnight bladder drainage on bladder function evaluated by urodynamics study, renal function estimated by SCr, eGFR and DMSA scan and on febrile urinary tract infections assessed by urinalysis and urine culture.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elkashef, Principal Investigator — Urology and Nephrology Center, Mansoura University, Egypt; Ahmed Abdelhalim, Study Director — Urology and Nephrology Center, Mansoura University, Egypt; Ashraf Hafez, Study Director — Urology and Nephrology Center, Mansoura University, Egypt; Mohamed Dawaba, Study Director — Urology and Nephrology Center, Mansoura University, Egypt
Locations (1):
- Urology and Nephrology Center, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: No